CLINICAL TRIAL: NCT02119494
Title: POPE-Study: Phenotypes Of COPD in Central and Eastern Europe Study
Brief Title: Phenotypes of COPD in Central and Eastern Europe
Acronym: POPE
Status: Completed | Type: Observational
Sponsor: Zuzana Zbožínková, M.Sc. (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Zuzana Zbožínková, M.Sc., project manager, Masaryk University
Organization: Masaryk University (Other)
Other Study IDs: 205.529
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; phenotypes; categories; stage; GOLD; treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the representation of COPD patients in terms of categories and phenotypes of the disease in selected countries in Central and Eastern Europe (CEE). The results of The POPE study will allow for evaluation of the differences in clinical approaches and treatment practices. The following countries are represented in The POPE study: Czech Republic, Slovakia, Austria, Poland, Hungary, Russia, Croatia, Serbia, Slovenia, Estonia, Latvia and Bulgaria.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a significant cause of morbidity and mortality in Europe and a major consumer of resources in both primary and secondary healthcare (1,2). Both clinical features of disease severity and quality of COPD patient care may have substantial influence on disease outcomes. Traditionally, COPD has been categorized using the FEV1 (forced expiratory volume at one second ) - based GOLD (The Global Initiative for Chronic Obstructive Lung Disease) classification . Other factors independently associated with survival include age, dyspnoea, health status, hyperinflation, gas exchange abnormalities, exacerbation frequency, exercise capacity, pulmonary hemodynamic, and nutritional status (3). Together these factors explain some of the existent heterogeneity within each GOLD stage in terms of symptoms, exacerbations, quality of life and exercise capacity (4).

Recently, interest has emerged for the identification of clinical COPD phenotypes, as defined by ''a single or combination of disease attributes that describe difference between individuals with COPD as they relate to clinically meaningful outcomes'' (5). Many previous studies have attempted to identify and quantify the prevalence of different phenotypes of COPD using populations of various sources, severities, and particularities. Yet there is no consensus on the number and definition of different phenotypes. However, there must be a compromise between the oversimplification of the term COPD as a definition that encompasses the entire spectrum of patients with incompletely reversible airflow obstruction caused largely by smoking and the complexity of considering each patient individually as an orphan disease.

The most frequently reported phenotypes are emphysema and chronic bronchitis, along with a subset of asthma sufferers. Recently, an extended list of proposed phenotypes have been proposed (6) including: (A) infrequent exacerbators with either chronic bronchitis or emphysema; (B) overlap COPD-asthma; (C) frequent exacerbators with emphysema predominant; and (D) frequent exacerbators with chronic bronchitis predominant. While there is consensus of substantial, but not complete, overlap among these phenotypes, the distribution of these phenotypes may differ widely between different countries and healthcare systems.

Thus, the objectives of this study are to better understand the patient characteristics and treatment patterns of those diagnosed with COPD between different CEE countries. Knowledge of this information may provide insight into the variability of phenotypes between different healthcare systems and may subsequently contribute to a better understanding of the factors associated with patient outcomes and have the potential to improve the care of COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 40 years
2. Clinical diagnosis of COPD with post-bronchodilator FEV1/FVC < 0.7
3. Smoking burden ≥ 10 pack-years in smokers (group A). Evidence of exposure to at least one other typical inhaled COPD risk factor: environmental tobacco smoke, professional exposures, etc. (group B) Each country will include 300 COPD subjects with positive history of smoking (at least 10 pack-years). Consecutive non-smokers with COPD can be enrolled above this limit. Institute for Biostatistics and Analyses, Masaryk University, Brno, The Czech Republic will analyze both COPD groups (A and B) separately
4. Stable disease for at least 4 weeks
5. Outpatient status
6. Informed Consent

Exclusion Criteria:

1. Exacerbation of COPD and/or instable co-morbid condition
2. Patient during hospital stay for whatever reason (lung or co-morbidities)
3. Patient is not able and willing to participate

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD who visit selected specialised pulmonology clinics in the given time period.
Sampling Method: Non-Probability Sample
Enrollment: 3504 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The distribution of COPD patients according to GOLD 2011 grades | 7 months
  The Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2011 classifies patients according to airflow limitation into four grades: GOLD1, Mild; GOLD 2, Moderate; GOLD 3, Severe; GOLD 4, Very severe
The distribution of COPD patients according to GOLD 2011 categories of risk (A. B, C, D) | 7 months

SECONDARY OUTCOMES:
The prevalence of various COPD phenotypes | 7 months
  The COPD phenotypes are: bronchitis, emphysema phenotype, frequent exacerbators, pulmonary cachexia, COPD and asthma overlap, and COPD and bronchiectasis overlap
The prevalence various medication prescription | 7 months
The prevalence of long term oxygen therapy use | 7 months
The prevalence of surgical treatments in COPD patients | 7 months
The use of body plethysmography, bronchodilator test, carbon monoxide diffusing capacity testing, bronchial challenge test and FeNO test in ambulatory care | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Arschang Valipour, Assoc. Prof., MD, PhD, Study Director — Vienna Hospital Association; Vladimir Koblizek, MD, Ph.D, Study Director — University Hospital Hradec Kralove; Ruzena Tkacova, Prof., MD, PhD, Study Director — Pavol Jozef Šafárik University in Košice; Neven Tudoric, Prof., MD, Ph.D, Study Director — University of Zagreb, Clinical Hospital Dubrava; Kyrill Zykov, MD, PhD, Study Director — Moscow State University of Medicine and Dentistry; Attila Somfay, Prof., MD, PhD, Study Director — University of Szeged, Faculty of Medicine, Dept. of Pulmonology; Adam Barczyk, MD, PhD, Study Director — Katedra i Klinika Pneumonologii, Śląski Uniwersytet Medyczny; Marc Miravitlles, Prof., MD, PhD, Study Director — Hospital Universitari Vall d'hebron Barcelona, Spain
Locations (81):
- Austria (5):
  - Department of Internal Medicine, University Innsbruck, Innsbruck
  - AKH Linz, Department of Pulmonary Medicine, Linz
  - SKA der PV Weyer/Enns, Mühlein
  - Pulmonary Rehabilitation Centre, Therme Wien, Vienna
  - Ludwig Boltzmann Institute, Vienna
- Bulgaria (4):
  - Clinic for pneumonology and phisiatry, UMHAT "Dr. Georgi Stranski", Pleven
  - Department of Respiratory Diseases, Medical University, Plovdiv
  - Pulmonary Diseases Clinic, Military Medical Academy, Sofia
  - Clinic of Pulmonology, MHAT "st. Marina", Varna
- Croatia (5):
  - Clinical Hospital, Osijek
  - University Hospital Centre, Rijeka
  - University Hospital Centre, Split
  - University Hospital Centre, Zagreb
  - University Hospital Dubrava, Zagreb
- Czechia (4):
  - Pulmonary Outpatient Clinic, University Hospital Hradec Králové, Hradec Králové
  - Plicní ambulance Karlovy Vary, Karlovy Vary
  - Plicní ambulance Ostrava Poruba, Ostrava
  - Plicní ambulance Teplice, Teplice
- Hungary (10):
  - Baja St. Rókus Hospital Patient Lung Care Institute, Baja
  - IZO PULM Health Service Ltd., Budapest
  - Újpest Non-Profit Health Care Services Ltd., Budapest
  - Csongrád County Hospital for Chest Diseases, Deszk
  - Medical Institution of Dr. Laszlo Romics Pulmonary Care, Érd
  - Elizabeth House Care Ltd., Gödöllő
  - St. Elizabeth Hospital Pulmonary Care Institute, Jászberény
  - Szabolcs-Szatmár-Bereg County Hospitals and University Teaching Hospital, Nyíregyháza
  - Federated Institutes of Health Institute of Pulmonary Care, Pécs
  - Szarvas Respiratory Ltd., Szarvas
- Latvia (19):
  - Health Centre Balvi, Balvi
  - Bauska Hospital, Bauska
  - Ambulatory Clinic Jelgava, Jelgava
  - Regional Hospital of Jekabpils, Jēkabpils
  - Ambulatory Clinic Dubulti, Jūrmala
  - Kuldīga Hospital, Kuldīga
  - Regional Hospital of Liepaja, Liepāja
  - Madona Hospital, Madona
  - Privat practice Viktorija Vevere, Rēzekne
  - Health Centre 4, Ltd, Riga
  - LU MPI Institute privat practice, Riga
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga 1st Hospital, Riga
  - Riga East Clinical University Hospital, In-patient Department "Centre of Tuberculosis and Lung Diseases, Riga
  - UniClinic, Riga
  - Health Centre, Talsi
  - rivat practice Ilona Uzbeka, Valka
  - Privat practice Dace Harasimjuka, Valmiera
  - Sia "Bini", Ventspils
- Poland (7):
  - Oddział Chorób Płuc i Niewydolności Oddychania, Kujawsko - Pomorskie; Centrum Pulmonologii w Bydgoszczy, Bydgoszcz
  - Klinika Alergologii i Pneumonologii, Uniwersyteckie Centrum Kliniczne, Szpital Gdańskiego Uniwersytetu Medycznego,, Gdansk
  - Oddział Chorób Płuc, Wojewódzkie Centrum Szpitalne Kotliny Jeleniogórskiej,, Jelenia Góra
  - Katedra i Klinika Pneumonologii, Śląski Uniwersytet Medyczny, Katowice
  - Szpital Uniwersytecki, Oddział Kliniczny Kliniki Pulmonologii, Krakow
  - Katedra i Klinika Pulmonologii, Alergologii i Onkologii Pulmonologicznej, Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Katedra i Klinika Chorób Wewnętrznych, Pneumonologii i Alergologii, Samodzielny Publiczny Centralny Szpital Kliniczny Warszawski Uniwersytet Medyczny,, Warsaw
- Russia (9):
  - State Budget Educational Institution of High Professional Education "Kazan State Medical University", Kazan'
  - I.M.Sechenov First Moscow State Medical University, University Hospital #1, Outpatient Department, Moscow
  - Moscow State City Clinical Hospital No. 24, Moscow
  - Moscow State University of Medicine and Dentistry named after A.I.Evdokimov, Moscow
  - Pulmonology Research Institute, Moscow
  - Clinic of Pulmonology of Scientific and Clinical Center of Interstitial and Orphan Lung Diseases, Saint Petersburg
  - GBOU VPO Samara State Medical University, Samara
  - Ufa State City Clinical Hospital, Ufa
  - Vladivostok Clinical Hospital No.1, Vladivostok
- Serbia (5):
  - Clinic for Pulmonary Diseases, Clinical Centre of Serbia, Belgrade
  - Municipal Institute for Lung Diseases and Tuberculosis, Belgrade
  - Clinic for Pulmonary Diseases, Clinical Centre Kragujevac, Kragujevac
  - Clinic for Pulmonary Diseases, Clinical Center of Nis, Niš
  - Institute for Pulmonary Diseases and TB, Clinical Centre Vojvodina, Novi Sad
- Slovakia (10):
  - FNsP F.D. Roosevelta, Banská Bystrica
  - NsP Sv. Jakuba, Bardejov
  - Klinika pneumológie a ftizeológie LF SZU a UNB,, Bratislava
  - Zdravotné stredisko Fedinova, Bratislava
  - Ambulancia pneumológie a ftizeológie, ZAPA JJ s.r.o.,, Levice
  - Klinika tubekulózy a respiračných chorôb JLF UK a UNM, Martin
  - Dionea, s.r.o., Nové Zámky
  - Pľúcna ambulancia, Poprad
  - NsP, Považská Bystrica
  - Zdravotné stredisko Rimava, Rimavská Sobota
- Slovenia (3):
  - Alveola, d.o.o., Maribor
  - Zdravstveni dom Murska Sobota, Murska Sobota
  - Bolnišnica Topolšica, Topolšica

REFERENCES:
- [Background] Gershon AS, Wang C, Wilton AS, Raut R, To T. Trends in chronic obstructive pulmonary disease prevalence, incidence, and mortality in ontario, Canada, 1996 to 2007: a population-based study. Arch Intern Med. 2010 Mar 22;170(6):560-5. doi: 10.1001/archinternmed.2010.17. PMID 20308643
- [Background] Menn P, Heinrich J, Huber RM, Jorres RA, John J, Karrasch S, Peters A, Schulz H, Holle R; KORA Study Group. Direct medical costs of COPD--an excess cost approach based on two population-based studies. Respir Med. 2012 Apr;106(4):540-8. doi: 10.1016/j.rmed.2011.10.013. Epub 2011 Nov 18. PMID 22100535
- [Background] Dolan S, Varkey B. Prognostic factors in chronic obstructive pulmonary disease. Curr Opin Pulm Med. 2005 Mar;11(2):149-52. doi: 10.1097/01.mcp.0000153548.36054.8f. PMID 15699788
- [Background] Agusti A, Calverley PM, Celli B, Coxson HO, Edwards LD, Lomas DA, MacNee W, Miller BE, Rennard S, Silverman EK, Tal-Singer R, Wouters E, Yates JC, Vestbo J; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) investigators. Characterisation of COPD heterogeneity in the ECLIPSE cohort. Respir Res. 2010 Sep 10;11(1):122. doi: 10.1186/1465-9921-11-122. PMID 20831787
- [Background] Han MK, Agusti A, Calverley PM, Celli BR, Criner G, Curtis JL, Fabbri LM, Goldin JG, Jones PW, Macnee W, Make BJ, Rabe KF, Rennard SI, Sciurba FC, Silverman EK, Vestbo J, Washko GR, Wouters EF, Martinez FJ. Chronic obstructive pulmonary disease phenotypes: the future of COPD. Am J Respir Crit Care Med. 2010 Sep 1;182(5):598-604. doi: 10.1164/rccm.200912-1843CC. Epub 2010 Jun 3. PMID 20522794
- [Background] Miravitlles M, Soler-Cataluna JJ, Calle M, Molina J, Almagro P, Quintano JA, Trigueros JA, Pinera P, Simon A, Riesco JA, Ancochea J, Soriano JB. A new approach to grading and treating COPD based on clinical phenotypes: summary of the Spanish COPD guidelines (GesEPOC). Prim Care Respir J. 2013 Mar;22(1):117-21. doi: 10.4104/pcrj.2013.00016. PMID 23443227
- [Derived] Miravitlles M, Koblizek V, Esquinas C, Milenkovic B, Barczyk A, Tkacova R, Somfay A, Zykov K, Tudoric N, Kostov K, Zbozinkova Z, Svoboda M, Sorli J, Krams A, Valipour A. Determinants of CAT (COPD Assessment Test) scores in a population of patients with COPD in central and Eastern Europe: The POPE study. Respir Med. 2019 Apr;150:141-148. doi: 10.1016/j.rmed.2019.03.007. Epub 2019 Mar 21. PMID 30961941
- [Derived] Tudoric N, Koblizek V, Miravitlles M, Valipour A, Milenkovic B, Barczyk A, Somfay A, Zykov K, Kostov K, Zbozinkova Z, Svoboda M, Sorli J, Krams A, Tkacova R. GOLD 2017 on the way to a phenotypic approach? Analysis from the Phenotypes of COPD in Central and Eastern Europe (POPE) Cohort. Eur Respir J. 2017 Apr 26;49(4):1602518. doi: 10.1183/13993003.02518-2016. Print 2017 Apr. No abstract available. PMID 28446560
- [Derived] Zbozinkova Z, Barczyk A, Tkacova R, Valipour A, Tudoric N, Zykov K, Somfay A, Miravitlles M, Koblizek V. POPE study: rationale and methodology of a study to phenotype patients with COPD in Central and Eastern Europe. Int J Chron Obstruct Pulmon Dis. 2016 Mar 22;11:611-22. doi: 10.2147/COPD.S88846. eCollection 2016. PMID 27042048